CLINICAL TRIAL: NCT01533532
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind Phase II Study of KLH-2109 in Patients With Endometriosis(2)
Brief Title: A Randomized, Placebo-controlled, Double-blind Study of KLH-2109 in Patients With Endometriosis (2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KLH1202
Record Dates: First submitted 2012-02-12; First posted 2012-02-15 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Endometriosis
Keywords: Gonadotropin-Releasing Hormone (GnRH) antagonist
MeSH Terms: conditions — Endometriosis | interventions — linzagolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- KLH-2109, low dose (Experimental)
  Interventions: Drug: KLH-2109
- KLH-2109, medium dose (Experimental)
  Interventions: Drug: KLH-2109
- KLH-2109, high dose (Experimental)
  Interventions: Drug: KLH-2109
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: KLH-2109
  Arms: KLH-2109, low dose
Drug: KLH-2109
  Arms: KLH-2109, medium dose
Drug: KLH-2109
  Arms: KLH-2109, high dose
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KLH-2109 in patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with endometriosis

Exclusion Criteria:

* Patients with clinically significant hepatic, renal, or cardiovascular dysfunction

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100

PRIMARY OUTCOMES:
The severity score of the pelvic pain | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuro Takei, Study Director — Clinical Development Dept.,Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Japan, Tokyo and Other Japanese City, Japan